CLINICAL TRIAL: NCT00574808
Title: Improved Delivery of Cardiovascular Preventive Care (IDOCC) Through Outreach Facilitation
Brief Title: Improved Delivery of Cardiovascular Care Through Outreach Facilitation
Acronym: IDOCC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: C. T. Lamont Primary Care Research Centre (Other)
Collaborators: Dept of Family Medicine, Faculty of Medicine, Hebrew University, Jerusalem, Israel (Other); Institute of Population Health, University of Ottawa (Other); Ottawa Heart Institute Research Corporation (Other); Ottawa Cardiovascular Centre (Unknown); Ottawa Regional Stroke Program (Unknown); Bruyère Health Research Institute. (Other); Champlain Primary Care Practices (Unknown)
Responsible Party: Principal Investigator, Dr. William Hogg, Dr., C. T. Lamont Primary Care Research Centre
Organization: Bruyère Health Research Institute. (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: IDOCC; 937200801
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Hypertension; Dyslipidemia; Diabetes; Chronic Kidney Disease; Cardiovascular Disease; Stroke; Transient Ischemic Attacks
Keywords: Primary care; Prevention of Cardiovascular Disease; Chronic Disease Management; Chronic Disease Prevention; Chronic Care Model; Outreach Facilitation
MeSH Terms: conditions — Hypertension; Dyslipidemias; Diabetes Mellitus; Renal Insufficiency, Chronic; Cardiovascular Diseases; Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): Outreach Facilitation implementing elements of the Chronic Care Model. The facilitators will provide hands on support to practices and help to implement tools and processes designed to incorporate evidence-based practice into the routine delivery of cardiovascular care. Specifically, they will a) assist with practice performance assessment, feedback, and consensus building towards goal setting, b) offer clinical, technical, organizational resources and practical advice, and c) provide encouragement to face and overcome the challenges of implementing system change.
  Interventions: Other: Outreach Facilitation implementing elements of the Chronic Care Model
- control (No Intervention): Baseline data before implementation of the program will serve as the control. Comparisons will be made between baseline and post-intervention within each divisions of primary care practices as well as between divisions (ie. baseline information from one division will serve as the control for another).

INTERVENTIONS:
Other: Outreach Facilitation implementing elements of the Chronic Care Model — An outreach facilitator helps the practice identify areas for improvement, set goals and targets, and agree on the processes needed to reach them in order to improve the care delivery within the practices. Each facilitator will be assigned up to 12 practice sites. The first year of program implementation will involve frequent (once every 3-4 weeks) visits to the practices. Afterwards, the intervention will move into a sustainability mode, during which the frequency of visits will decrease to one every 6-8 weeks during the second year, and one every 12-15 weeks during the third year and thereafter. After the first year of program implementation, each facilitator will be able to take on 12 new practices during the second year, while still being able to sustain contact with the previous 12 practices. Similarly, in the third year, another set of 12 practices will begin the "intense" phase of program implementation.
  Arms: intervention

SUMMARY:
The aim of the proposed study is to implement and evaluate Outreach Facilitation as a means to increase the uptake of evidence-based practice for secondary prevention and management of patients with established CVD and cardiovascular risk factors, in primary care practices throughout the Champlain LHIN. This initiative centers on the use of an Outreach Facilitation Model, in which skilled health professionals known as facilitators (Practice Change Consultants) serve as an expert resource to primary care practices in three areas: a) practice performance assessment, feedback, and consensus building towards goal setting and implementation; b) clinical, technical, organizational resources and practical advice; and c) encouragement to face and move through the challenges associated with implementing system change.

DETAILED DESCRIPTION:
General practice visits can provide a unique opportunity to identify and treat individuals with or at risk for CVD. We plan to test implementation of system changes using nurse facilitation in the organization of primary care practices to enhance daily adoption by the practice staff of evidence-based guidelines and prevention strategies that can lead to better patient care.

Specifically, we will:

i) Establish an Outreach Facilitation program in primary care practices throughout the Champlain District to improve the secondary prevention and management of cardiovascular disease in the primary care setting. The program will assist the practices (Champlain CVD Prevention Network) with implementation of evidence-based guidelines (Champlain Primary Care CVD Prevention Guidelines) by targeting the following risk factors:

* Hypertension
* Dyslipidemia
* Diabetes
* Chronic Kidney Disease
* Smoking
* Obesity
* Physical Inactivity

ii) Rigorously evaluate this program's efficacy and cost effectiveness

Hypotheses

Implementation of the outreach facilitation program for CVD prevention and management will improve: i) the processes of cardiovascular health related care delivery by primary care practitioners in the Champlain LHIN, and ii) the clinical outcomes for patients with established CVD and those at high cardiovascular risk. The improvements will be evident on the comparisons of the pre- to post-implementation performance within the participating practices, and on the between practice comparisons of performance in those randomized to begin the program earlier with those randomized to begin it later.

Design

We will use a "stepped wedge" design where the outreach facilitation program will be rolled-out sequentially to the trial participants, in geographic regions chosen by random order, over a number of equally spaced time intervals during the 5 year program implementation period.

To allow for the sequential roll-out of the program, the Champlain LHIN has been divided into 9 smaller geographic regions, referred to from now on as "divisions", using GIS mapping technology. The order in which these divisions begin the program has been randomized, but stratified by the west/central/and east location within the LHIN, so that each division per stratum will have the same probability of beginning the program at any specific time.

There will be 4 data collection points throughout the 5-year implementation period. In the analysis, the data points before program implementation (the baseline section of the wedge) will be compared to the data points after the program begun (the implementation section of the wedge) both within and between the divisions. The multiple baseline data obtained for those divisions randomized to begin the program later than others will allow for underlying temporal changes to be considered as a variable in data analysis in order to determine, for example, whether any secular changes had an impact on effectiveness of the program.

Impact Evaluation

To measure the population-level impact of the program we will collaborate with the Institute for Clinical Evaluative Sciences (ICES). Specifically, we will evaluate the regional impact of the program on cardiovascular health by linking participating doctors with provincial administrative databases from ICES to determine the rates of CVD-related hospitalization and emergency department visits, mortality and morbidity, and drug prescription patterns for hypertension, lipid control, and other vascular protective agents.

In addition, we will measure the success of the program at the level of the primary care practice through a qualitative assessment of the following aspects of program implementation:

* the impact of the intervention on physicians, associated staff and patients
* the resources and activities required to implement the intervention and the extent to which it was implemented as intended
* the factors which contributed to success or which introduce barriers to success

Satisfaction with the program will be evaluated at the level of the physician, practice staff, and the facilitators.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 40 years of age, who meet at least one of the following criteria:

  1. have established cardiovascular disease: Coronary Artery Disease, Cerebrovascular disease (documented stroke and/or TIA), and Peripheral Vascular Disease;
  2. have Diabetes Mellitus;
  3. have Chronic Kidney Disease ;
  4. are at high risk for CVD based on a presence of at least three of the following established cardiovascular risk factors: age (males ≥ 45, females ≥ 55), smoker status, hypertension, and dyslipidemia.
* No restrictions will be imposed on the recruitment process; all practices in the region will be eligible to participate.

Exclusion Criteria:

* see above

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2007-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Quality of care process index = ∑ of recommended services received by patient/ ∑ of the recommended services for which the patient was eligible | 5 years

SECONDARY OUTCOMES:
Quality of care outcome index = ∑ of recommended targets reached / ∑ of the number of targets for which the patient is eligible based on the number of conditions suffered by the patient | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clare E Liddy, MD, MSc, Principal Investigator — University of Ottawa; William Hogg, MD, MSc, Principal Investigator — University of Ottawa
Locations (1):
- Elisabeth Bruyere Health Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Lemelin J, Hogg W, Baskerville N. Evidence to action: a tailored multifaceted approach to changing family physician practice patterns and improving preventive care. CMAJ. 2001 Mar 20;164(6):757-63. PMID 11276541
- [Background] Baskerville NB, Hogg W, Lemelin J. Process evaluation of a tailored multifaceted approach to changing family physician practice patterns improving preventive care. J Fam Pract. 2001 Mar;50(3):W242-9. PMID 11252222
- [Background] Hogg W, Baskerville N, Lemelin J. Cost savings associated with improving appropriate and reducing inappropriate preventive care: cost-consequences analysis. BMC Health Serv Res. 2005 Mar 9;5(1):20. doi: 10.1186/1472-6963-5-20. PMID 15755330
- [Derived] Liddy C, Rowan M, Valiquette-Tessier SC, Drosinis P, Crowe L, Hogg W. Improved Delivery of Cardiovascular Care (IDOCC): Findings from Narrative Reports by Practice Facilitators. Prev Med Rep. 2016 Dec 23;5:214-219. doi: 10.1016/j.pmedr.2016.12.018. eCollection 2017 Mar. PMID 28271017
- [Derived] Deri Armstrong C, Taljaard M, Hogg W, Mark AE, Liddy C. Practice facilitation for improving cardiovascular care: secondary evaluation of a stepped wedge cluster randomized controlled trial using population-based administrative data. Trials. 2016 Sep 5;17(1):434. doi: 10.1186/s13063-016-1547-2. PMID 27596224
- [Derived] Liddy C, Hogg W, Singh J, Taljaard M, Russell G, Deri Armstrong C, Akbari A, Dahrouge S, Grimshaw JM. A real-world stepped wedge cluster randomized trial of practice facilitation to improve cardiovascular care. Implement Sci. 2015 Oct 28;10:150. doi: 10.1186/s13012-015-0341-y. PMID 26510577
- [Derived] Liddy C, Singh J, Hogg W, Dahrouge S, Deri-Armstrong C, Russell G, Taljaard M, Akbari A, Wells G. Quality of cardiovascular disease care in Ontario, Canada: missed opportunities for prevention - a cross sectional study. BMC Cardiovasc Disord. 2012 Sep 12;12:74. doi: 10.1186/1471-2261-12-74. PMID 22970753
- [Derived] Liddy C, Singh J, Hogg W, Dahrouge S, Taljaard M. Comparison of primary care models in the prevention of cardiovascular disease - a cross sectional study. BMC Fam Pract. 2011 Oct 18;12:114. doi: 10.1186/1471-2296-12-114. PMID 22008366
- [Derived] Liddy C, Hogg W, Russell G, Wells G, Armstrong CD, Akbari A, Dahrouge S, Taljaard M, Mayo-Bruinsma L, Singh J, Cornett A. Improved delivery of cardiovascular care (IDOCC) through outreach facilitation: study protocol and implementation details of a cluster randomized controlled trial in primary care. Implement Sci. 2011 Sep 27;6:110. doi: 10.1186/1748-5908-6-110. PMID 21952084